CLINICAL TRIAL: NCT06465888
Title: Evaluating the Influence of Egg Nutrients on Visual Cognitive Performance in Older Adults: A Randomized Controlled Trial
Brief Title: Influence of Eggs on Cognitive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Egg Nutrition Center (Other)
Responsible Party: Principal Investigator, Steven E.Riechman, PhD, MPH, Associate Professor, Texas A&M University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: IRB2017-0379D
Record Dates: First submitted 2024-06-13; First posted 2024-06-20 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Function
Keywords: lutein; zeaxanthin; macular pigment optical density (MPOD); macular pigment; eggs; cognition; cognitive performance
MeSH Terms: interventions — Egg White; Egg Yolk

STUDY DESIGN:
Intervention Model Description: This is a 30-day study. Serum analysis and diagnostic testing will be conducted at baseline. Participants will be randomly assigned to a no-egg control or one of the following dietary treatment groups: 4 large egg whites daily; 2 large whole eggs daily; 2 large whole omega-3 fortified eggs daily; or 4 large egg yolks daily. Participants will be asked to follow their routine food and beverage intake other than the assigned dietary treatment guidelines. Fifteen food logs will be completed. The last two weeks will include 15 Neurotracker 3-D cognitive training sessions over 10 days with diagnostic measures, physical activity, and sleep patterns recorded. Serum blood draw at day 30.
Who Masked: Participant
Masking Description: Brand name of eggs on cartons will be covered so participants will not know which eggs they were eating.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- No-Egg Control Group (No Intervention): The No-Egg Control group will not eat eggs or foods with eggs being one of the primary components of the food for 30 days.
- Egg White Group (Active Comparator): Participants will eat four egg whites/day for 30 days. Participants will be given a specified number of Kieke eggs to last them until their next appointment. They will be asked to eat no other eggs than whites from the eggs given to them and to return cartons with any leftover eggs.
  Interventions: Other: egg whites
- Whole Egg Group (Active Comparator): Participants will eat two whole eggs/day for 30 days. Participants will be given a specified number of Kieke eggs to last them until their next appointment. They will be asked to eat no other eggs than the eggs given to them and to return cartons with any leftover eggs.
  Interventions: Other: whole eggs
- Whole Omega-3 Egg Group (Active Comparator): Participants will eat two Christopher Farms whole omega-3 eggs/day for 30 days. Participants will be given a specified number of Christopher Farm eggs that will last them until their next appointment. They will be asked to eat no other eggs than the two from the eggs given to them and to return cartons with any leftover eggs.
  Interventions: Other: Omega-3 eggs
- Egg Yolk Group (Active Comparator): Participants will eat four egg yolks/day for 30 days. Participants will be given a specified number of Kieke eggs to last them until their next appointment. They will be asked to eat no other eggs than the yolks from the eggs given to them and to return cartons with any leftover eggs.
  Interventions: Other: egg yolk

INTERVENTIONS:
Other: egg whites — Participants will eat four egg whites daily for the 4-week study
  Arms: Egg White Group
Other: whole eggs — Participants will eat two eggs daily for the 4-week study
  Arms: Whole Egg Group
Other: Omega-3 eggs — Participants will eat two Christopher Farms omega-3 fortified eggs daily for the 4-week study.
  Arms: Whole Omega-3 Egg Group
Other: egg yolk — Participants will eat four egg yolks daily for the 4-week study
  Arms: Egg Yolk Group

SUMMARY:
This clinical trial aims to evaluate the nutrients in eggs in healthy adult's cognitive performance. The main questions it aims to answer are:

* How do the nutrients in eggs impact visual cognitive performance (VCP) in generally healthy older individuals?
* Will omega-3 fatty acids in eggs improve VCP in generally healthy older individuals?

Participants will be randomly placed in one of five dietary treatment groups, including four egg whites, two whole regular eggs, two whole omega-3 fortified eggs, four egg yolks, and a no-egg control. Blood will be drawn at baseline. During the first two weeks, participants will eat assigned eggs, consume their usual diet other than the eggs, and keep five food logs. Cognitive performance testing will start on day 15 and be measured over a 10-day period using the Neurotracker (NT) 3-D program. Data on ancillary factors influencing outcomes will be collected, and food will be logged on each NT training day. Blood will be drawn at the end of the study and compared with baseline levels.

DETAILED DESCRIPTION:
Generally, healthy males or 2 years post-menopausal females between 50 and 75 years old will be recruited for this study. Potential subjects will communicate interest to researchers, and a standardized email with a consent form will be sent to persons of interest. Prospective participants will complete a preliminary questionnaire evaluating visual health to confirm inclusion criteria met, a study ID will be assigned. subjects will be randomly placed in a control group or one of four intervention groups: four egg whites, two whole regular eggs, two whole omega-3 eggs, and four egg yolks. Eggs will be provided to subjects based on their treatment groups; egg distribution will occur on days 1 and 15. Fifteen days of food logs, five days during the first 14 days of the study, and ten days of food logs each day the subjects train on the Neurotracker software. Food logs will be analyzed using Nutribase software.

Two weeks after the commencement of the study (Day 15), cognitive performance testing will begin. This testing will be conducted over a 10-day period, consisting of 15 training sessions. The Neurotracker (NT) 3-D program will be used for these sessions. On each NT training day, a daily data questionnaire will be used to collect data on ancillary factors that may influence the outcomes of the study.

Blood will be drawn at baseline, on day 15, and at the end of the study. Average nutrient intake and dietary patterns, baseline plasma draws, rate of change, and maximal performance on the NT software will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and post-menopausal women who are age 50 to 75 years

Exclusion Criteria:

* Taking supplements with >6 mg L and/or >2 mg Z two months before the study
* Self-reported diagnosis of age-related macular degeneration, diabetic retinopathy, glaucoma, or other eye conditions that may negatively impact visual cognitive performance

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Cognitive performance | 15 cognitive sessions within 10 days over 2 week period
  Neurotracker 3-Dimensional software used to measure cognitive performance. Subjects performed 20 trials within a single training session obtaining a "speed threshold," (ST) the level at which the participant correctly tracked and selected the correct objects 50% of the time. The final ST for each training session and the progression over 15 sessions were the primary determinants of cognitive performance.
Nutrient Intake (Lutein and Zeaxanthin) | Through study completion which may take up to 2 years.
  Serum will be drawn and analyzed for lutein and zeaxanthin content

SECONDARY OUTCOMES:
Serum Lipid Levels | Through study completion which may take up to 2 years.
  Serum will be drawn and analyzed for lipoprotein subfractions

CONTACTS AND LOCATIONS:
Overall Officials: Steven E. Riechman, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Gilchrist Building, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No